CLINICAL TRIAL: NCT05930886
Title: Focus Groups to Optimize Research Methodology in a Multinutrient Study of Racially and Ethnically Diverse Children With ADHD and Emotional Dysregulation
Brief Title: Focus Groups in Ethnically and Racially Diverse Families
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeanette Johnstone, Assistant Professor, Oregon Health and Science University
Other Study IDs: 00024335
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Emotional Dysfunction; Irritable Mood
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hispanic Community: 15 adult parents/caregivers self-identified as Hispanic
  Interventions: Other: Focus Group
- Black/African American Community: 15 adult parents/caregivers self-identified as Black/African American
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Black or Hispanic/Latino parents, caregivers or family members of children with ADHD symptoms and/or emotional dysregulation, will discuss: (1) impact of child's mental health, treatments, care received; (2) perceived and actual barriers to future study participation, including discussion about acceptability of bio-specimen collection methods for urine and blood. Each group will comprise individuals who self-identify as Hispanic/Latino, Black, or mixed race. Groups are anticipated to comprise individuals who identify with one or the the other race/ethnicity in order to create space to hear perspectives that may differ between these broadly defined groups.

SUMMARY:
Focus groups to identify treatment needs and barriers to participation in the planned multinutrient study among racially and ethnically diverse (Black and Hispanic) communities.

DETAILED DESCRIPTION:
Focus group purpose is to understand parents' priorities regarding their child's mental health, and facilitators or barriers to research participation generally, with inquiry about CIH intervention use, and the multinutrient feasibility study specifically. Researchers will engage Black and Hispanic families in focus groups to discuss mental health priorities related to their children, and real or perceived barriers to engagement in research studies. The feedback will inform the final design and recruitment for the multinutrient feasibility study in Black and Hispanic populations. One group will comprise individuals who self-identify as Hispanic, another, as Black, in order to create space to hear perspectives that may differ between broadly defined groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult parents/caregivers self-identified as Black or Hispanic/Latino
* With a family member 6-18 years old with suspected ADHD and/or emotional dysregulation, or provide care for, or teach someone who meets these criteria
* Who have sought or are interested in treatment
* Willing to discuss child's mental health care needs and provide feedback regarding feasibility study
* Able to attend focus groups in person
* Able to communicate in English or Spanish
* Agree to focus group session audio recording

Exclusion Criteria:

* Unwilling to be recorded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community samples of Portland, Oregon individuals who self-identify as Hispanic/Latino/a for one focus group and Black/African American for another.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-04 (Estimated)

PRIMARY OUTCOMES:
Input and Feedback on Proposed Feasibility Study | Baseline
  Purpose is understanding
  1. Parents' priorities regarding their child's mental health
  2. Facilitators or barriers to research participation generally
  3. Parent input on planned study specifically
  4. Specific recommendations for modifying the future feasibility study design
  5. Previous CIH intervention use

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Johnstone, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States